CLINICAL TRIAL: NCT01542398
Title: Title: Is a Family-based, Life Skills Focused Intervention Effective in Reducing Psychological Distress and Stigma and Improving Inter-personal Relations and Functioning Among Former LRA Abductees and Other War-affected Children in Their Community in Dungu, the Democratic Republic of Congo?
Brief Title: A Family-based, Resilience-focused Intervention for War-affected Communities in North-eastern Democratic Republic of Congo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Discover the Journey (Unknown)
Responsible Party: Principal Investigator, Paul O'Callaghan, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREC 06-2012
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-06

CONDITIONS: Psychological Distress
Keywords: community-based; war-affected; psychosocial support; family-focused; psychological distress; adolescents; Democratic Republic of Congo; family functioning; community functioning; daily functioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-Focused Psychosocial Intervention (Experimental): Intervention Group
  Interventions: Behavioral: Family-Focused, Community-Based, Resilience-Targetting Psychosocial Intervention
- Waiting List Control (No Intervention)

INTERVENTIONS:
Behavioral: Family-Focused, Community-Based, Resilience-Targetting Psychosocial Intervention — A 12-module manualised intervention focusing on reducing psychological distress, improving family and community functioning and boosting daily functioning of adolescents through the use of Mobile Cinema Screenings and task-based, participatory, group-sessions
  Arms: Family-Focused Psychosocial Intervention

SUMMARY:
The main research question of the study is whether a family-based, life-skills focused psychosocial intervention is effective in reducing psychological distress and stigma and improving inter-personal relations and functioning among war-affected children in the Democratic Republic of Congo.

ELIGIBILITY:
Inclusion Criteria:

* War-affected
* eastern Democratic Republic of Congo
* Formerly abducted child or vulnerable child

Exclusion Criteria:

* severe/violent behavioural problems
* severe learning difficulties

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciarán Shannon, BA, MA, DClin, Study Director — British Psychological Society (Chartered Clinical Psychologist)
Locations (1):
- Dungu, Dungu, Haut-Uele, Republic of the Congo

REFERENCES:
- [Derived] O'Callaghan P, Branham L, Shannon C, Betancourt TS, Dempster M, McMullen J. A pilot study of a family focused, psychosocial intervention with war-exposed youth at risk of attack and abduction in north-eastern Democratic Republic of Congo. Child Abuse Negl. 2014 Jul;38(7):1197-207. doi: 10.1016/j.chiabu.2014.02.004. Epub 2014 Mar 15. PMID 24636358

RESULTS

PARTICIPANT FLOW:
Groups:
- Family-Focused Psychosocial Intervention: Intervention Group
  Family-Focused, Community-Based, Resilience-Targetting Psychosocial Intervention: An 8-module manualised intervention focusing on reducing psychological distress, improving family and community functioning and boosting daily functioning of adolescents through the use of Mobile Cinema Screenings and task-based, participatory, group-sessions
- Waiting List Control Group: Waiting List Control Group of Adolescents who received the intervention once it was shown to be effective for the Intervention Group
Period: Overall Study
Arm/Group | Family-Focused Psychosocial Intervention | Waiting List Control Group
Started | 79 | 80
Post-Intervention Assessment | 78 | 80
Completed | 71 | 67
Not Completed | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family-Focused Psychosocial Intervention | Waiting List Control | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.16 (2.85) | 13.76 (2.76) | 13.42 (2.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 43 | 45 | 88
Region of Enrollment [Number; unit: participants]
  Congo | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Post-traumatic Stress Reaction Symptoms Among Participants
Description: To assess post-traumatic stress reaction symptoms the 8-item Impact of Events Scale (CRIES-8) was used (Yule, 1997). Respondents indicating how frequently they experience a symptom on a 4-point Likert scale (0, 1, 2, 3). Thus the minimum score was 0 while the maximum score was 24. A high score indicates a high level of post-traumatic stress symptoms. This 8-item CRIES, which was designed for children over 7 years of age, has an identical factor structure to the 22-item version (Yule, 1997) which was previously validated with a sample of 1,046 war-affected adolescents in the eastern Democratic Republic of Congo (Mels, Derluyn, Broekaert & Rosseel, 2010) (internal reliability range: 0·79 to 0·84; Cronbach's alpha for the total scale: 0·93). In the current study, internal consistency was 0·557.
Time Frame: 1-week before intervention, 3-weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-Focused Psychosocial Intervention | Waiting List Control Group
Number analyzed (Participants) | 79 | 80
units on a scale
  Pre-Intervention Mean Scores | 11.79 (5.28) | 11.80 (5.56)
  Post-Intervention Mean Scores | 12.17 (5.70) | 10.03 (4.76)

2. Secondary Outcome: African Youth Psychosocial Assessment Inventory - Depression and Anxiety Subscales
Description: Internalising symptoms were assessed using the African Youth Psychosocial Assessment Instrument (AYPA) (Betancourt et al., 2009).This 17 item Likert (0 = minimum, 51 = maximum) measure was developed in northern Uganda after extensive qualitative consultation with young people, caregivers and mental health workers. A high score on the AYPA indicates a high level of internalizing symptoms. It is the only African developed, validated questionnaire available, had been used in separate studies with war-affected children in the DR Congo (McMullen et al., 2013; O'Callaghan, McMullen, Shannon, Rafferty & Black; 2013) and includes symptoms of distress which do not appear in Western-developed measures (e.g. muttering to oneself, feeling pain in your heart, sitting with your head in your hand etc.). Test-retest reliability (carried out with a subset of 30 participants) for the AYPA was 0·91, inter-rater reliability was 0·58 (n = 26) and internal consistency was 0·787 (internalising symptoms).
Time Frame: pre-intervention, 3 weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-Focused Psychosocial Intervention | Waiting List Control
Number analyzed (Participants) | 79 | 80
units on a scale
  Pre-Intervention Scores | 14.88 (7.07) | 13.53 (6.19)
  3 week Post-Intervention Scores | 12.09 (6.26) | 11.57 (5.36)

ADVERSE EVENTS:
Time Frame: Participants were informally monitored (through thrice weekly check-ins with the village leaders who were supporting the intervention) to ensure that the study intervention was not causing harm or resulting in Adverse Events for people in either the intervention or waiting-list control group. No Adverse Events were reported to the team during the duration of the study or in the study month follow-up.
Description: Although all participants faces a real and concerning threat of abduction by rebel units operating in the area, during the study no abductions of participants took place and the two villages where the interventions occurred were not attacked. It must also be stated that although these were Serious Adverse Risks being faced by participants these risks were not created by the study and participants were free to leave their villages at any time, should they feel that this was necessary.
Arm/Group | Intervention Group | Waiting List Control Group
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 0/79 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No